CLINICAL TRIAL: NCT05208034
Title: Treatment Success With Two Doses of Methotrexate vs Single Dose of Methotrexate in Ectopic Tubal Pregnancy
Brief Title: Medical Treatment in Ectopic Tubal Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nishtar Medical University (Other)
Responsible Party: Principal Investigator, Rashida Parveen, Consultant Gynecologist, Nishtar Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NishtarMU12
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Ectopic Pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Methotrexate

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single-dose group (No Intervention): Women in single-dose group were administered a single-dose of intramuscular methotrexate as 50 mg/m2 on day-zero (the start of treatment).
- two-dose group (Experimental): Women allocated to two-dose group were administered intramuscular methotrexate as 50mg/m2 at day-zero and 7 while measurement of β-hCG was ordered at day-14.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Two-doses of intramuscular methotrexate as 50mg/m2.. One at at day-zero and 2nd at day 7.
  Arms: two-dose group

SUMMARY:
Ectopic pregnancy (EP) is estimated to be responsible for approximately 20% of all pregnancy-related mortality and 46% early pregnancy mortality.1 Hemodynamically stable women with EP are frequently managed with methotrexate (MTX) while multiple protocols like fixed multiple doses, single-dose as well as two-dose regimens have been in practice for treating EP, but no consensus exists regarding the optimum dosage regimen.

DETAILED DESCRIPTION:
Literature reports multiple dosage regimens of MTX to be associated with increased rates of side effects. Single dose protocol has good compliance and fewer side effects but is linked with lower success rates in comparison to multiple dose protocols.

A new treatment protocol involving "two-doses" of MTX for medical management of EP was introduced in 2007 but most of the research conducted so far has been retrospective in nature and limitations in study designs. No such study in recent years has been done in Pakistan to compare the success and safety of single-dose and two-dose MTX protocols so this study was planned to compare the success rates and safety of two-doses of MTX versus single dose of MTX in tubal EP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of tubal ectopic pregnancy.
* Pre-treatment beta-human chorionic gonadotrophin (β-hCG) level below 1500 mIU/ml.
* Gestational sac with largest diameter as 4cm.
* Willing to take methotrexate treatment.
* Willing to follow up.

Exclusion Criteria:

* Heterotrophic pregnancy
* Persistent tubal pregnancy
* Embryonic cardiac motion
* Suspected tubal rupture
* Past history of harmful effects of methotrexate treatment on organ functions.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
success rate | 4-14 days
  In single-dose group,β-hCG levels were measured at day-4 and 7 and if β-hCG decreased >15% between day-4 and day-7, the treatment was labeled successful.
  In two-dose group, in case 15% reduction in β-hCG level was observed at day-14, the treatment was labeled as success.

SECONDARY OUTCOMES:
frequency of Side-effects of treatment | 1-14 days
  monitoring for the side effects during the treatment duration
β-hCG Resolution Time | 1-14 days
  Time taken for β-hcg resolution to reduce below 15%

CONTACTS AND LOCATIONS:
Overall Officials: Rashida Parveen, FCPS, Principal Investigator — Nishtar Medical University
Locations (1):
- Nishtar Medical University Hospital, Multan Khurd, Pu, Pakistan

IPD SHARING:
Plan to Share IPD: No